CLINICAL TRIAL: NCT04645615
Title: European CURE-AF Study - Concomitant Utilization of Radiofrequency Energy for Atrial Fibrillation
Brief Title: European CURE-AF Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: European CURE-AF Study
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CURE AF (Experimental)
  Interventions: Device: Cardioblate surgical ablation system; Procedure: Surgical RF Ablation

INTERVENTIONS:
Device: Cardioblate surgical ablation system — This investigation is a prospective, non-randomized multicenter clinical trial evaluating the outcome of patients with AF requiring concomitant open heart surgery plus the Cardioblate Surgical Ablation System using the modified Maze III procedure. The trial population includes patients requiring valve replacements or repairs, atrial septal defect (ASD) repairs, patent foramen ovale (PFO) closure or coronary artery bypass grafts (CABG) procedures.
Procedure: Surgical RF Ablation — This investigation is a prospective, nonrandomized multicenter clinical trial evaluating the outcome of patients with AF requiring concomitant open heart surgery plus the Cardioblate Surgical Ablation System using the modified Maze III procedure. The trial population includes patients requiring valve replacements or repairs, atrial septal defect (ASD) repairs, patent foramen ovale (PFO) closure or coronary artery bypass grafts (CABG) procedures.

SUMMARY:
A prospective, non-randomized, multi-center clinical trial. The patient population includes patients with permanent or persistent AF requiring valve replacements or repairs, ASD repairs, PFO closure or coronary artery bypass grafts (CABG) procedures. Patients are not allowed to have had previous atrial ablation, AV-nodal ablation, or surgical Maze procedure.

DETAILED DESCRIPTION:
The Cardioblate Surgical Ablation System is cleared in Canada and Europe for ablation of cardiac tissue for the treatment of cardiac arrhythmias. In the United States, the Cardioblate bipolar is approved for soft tissue ablation, while the Cardioblate Pen is approved for cardiac tissue ablation. The purpose of the clinical study is to obtain a labeling claim for the US market that the Cardioblate Surgical Ablation System can be used for ablation of cardiac tissue in the treatment of cardiac arrhythmias such as atrial fibrillation among permanent and persistent AF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be enrolled in the study:

  1. Documented history of AF a For inclusion in permanent AF arm: Patients must have a documented history of permanent AF (cardioversion failure) as defined by the ACC/AHA/ESC Guidelines; Documentation of AF must include one or more chart references to AF and/or one or more ECG's with AF prior to the patient's surgery. Other supporting information could include references to cardioversion attempts using either drugs or electrical shock. b For inclusion in persistent AF arm: Patients must have a documented history of persistent AF as defined by the ACC/AHA/ESC Guidelines: characterized as episodes of non-self-terminating atrial fibrillation that usually lasts more than 7 days
  2. Concomitant indication (other than AF) for open-heart surgery for one or more of the following:

a Mitral valve repair or replacement, b Aortic valve repair or replacement, c Tricuspid valve repair or replacement, d ASD repair, e PFO closure, or f CABG procedures; 3 Able to take the anticoagulant warfarin or other ACC/AHA/ESC-recommended anticoagulant medication; 4 Greater than or equal to 18 years of age; 5 Able and willing to comply with study requirements by signing a Patient Informed Consent form.

Exclusion Criteria:

* Patients who meet any of the following criteria may not be enrolled in the study:

  1 Wolff-Parkinson-White syndrome, 2 NYHA functional class = IV, 3 Left ventricular ejection fraction ≤ 30%, 4 Left atrial diameter > 7.0 cm, 5. Need for emergent cardiac surgery (i.e. cardiogenic shock) or redo open heart surgery, 6 Preoperative need for an intra-aortic balloon pump or intravenous inotropes, 7 Previous atrial ablation, AV-nodal ablation, or surgical Maze procedure, 8 Contraindication for anticoagulation therapy, 9 Current diagnosis of active systemic infection, 10 Renal failure requiring dialysis or hepatic failure, 11 Documented myocardial infarction 6 weeks prior to study enrollment, 12 Life expectancy of less than one year, or 13 Pregnancy or desire to be pregnant within 12-months of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-06-19 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2013-07-10 (Actual)

PRIMARY OUTCOMES:
Permanent AF Arm | 24-hour Holter recording at 6 months follow-up
  Primary efficacy endpoint- The percent of patients free of AF, off Class I or III antiarrhythmic drugs and not having received additional ablation therapy, as determined by a 24-hour Holter recording at 6 months follow-up.
Persistent AF Arm | 24-hour Holter recording at 9 months follow-up.
  The percent of patients free of AF, off Class I or III antiarrhythmic drugs and not having received additional ablation therapy, as determined by a 24-hour Holter recording at 9 months follow-up.

SECONDARY OUTCOMES:
Permanent AF Arm | 24 hours
  Secondary efficacy endpoints - 24-hour Holter recording, b) improvement in left ventricular ejection fraction and c) left atrial transport function as evidenced by the presence of an A wave at 6 months follow-up.
Persistent AF Arm | 24-hour Holter recording at 9 months follow-up.
  Secondary efficacy endpoints - a) The percent of patients free of AF, regardless of Class I or III antiarrhythmic drug use and not having received additional ablation therapy, as determined by a 24-hour Holter recording, b) improvement in left ventricular ejection fraction and c) left atrial transport function as evidenced by the presence of an A wave at 9 months follow-up.

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (2):
  - Kerckhoff Clinic - Department of Thoracic & Cardiovascular Surgery, Bad Nauheim, Beneke Str. 2-8
  - Heart Center Cottbus - Department of Cardiac Surgery, Cottbus, Leipziger Strasse 50
- Norway (2):
  - St. Elizabeth Heart Center - Department of Cardiothoracic Surgery, Trondheim, Hans Nissens Gate 3
  - Haukeland University Hospital - Department of Cardiothoracic Surgery, Bergen, Jonas Liesvei 65
- Public Central Teaching Hospital - Department of Cardiac Surgery, Warsaw, Ul. Banacha 1a, Poland